CLINICAL TRIAL: NCT01895075
Title: Evaluation of the Effectiveness of Inhaled Budesonide for Non-ventilated Infants at High Risk of Bronchopulmonary Dysplasia: the i-BUD Pilot Study
Brief Title: Inhaled Budesonide for Non-ventilated Infants at High Risk of Bronchopulmonary Dysplasia: the i-BUD Pilot Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Dr. Michael Dunn (Other)
Responsible Party: Sponsor-Investigator, Dr. Michael Dunn, Staff neonatologist, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001-2013; CTRL # 165648 (Other: Health Canada)
Record Dates: First submitted 2013-06-25; First posted 2013-07-10 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Budesonide; Inhalation; Premature infants
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Respiratory Aspiration; Premature Birth | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaled budesonide (Experimental): Inhaled budesonide 1mg/dose (2ml) three tid
  Interventions: Drug: Inhaled budesonide
- Normal saline (Placebo Comparator): Normal saline inhalation 2ml tid
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Inhaled budesonide — Inhaled budesonide 1 mg tid until 36 weeks' corrected gestational age or fully weaned from supplemental oxygen and respiratory support (CPAP or high flow nasal canula)
  Other Names: PULMICORT® NEBUAMP®
  Arms: Inhaled budesonide
Drug: Normal saline — 2 ml normal saline by inhalation
  Other Names: Placebo
  Arms: Normal saline

SUMMARY:
Bronchopulmonary dysplasia (BPD) is one of the most important morbidities of preterm infants with a high incidence and significant impact on resource utilization and long-term outcome. Systemic corticosteroids have been shown to be effective in the prevention of BPD through their potent anti-inflammatory effects but there are serious concerns on their potential detrimental effects on neurodevelopment of infants. In contrast, inhaled corticosteroids administered to ventilated infants are thought to be safer due to their topical effect but have not been shown to improve outcomes including BPD. To date, there have been few studies evaluating the effect of inhaled corticosteroids administered to non-ventilated infants for the prevention of BPD. Hence, we are conducting a double-blind randomized controlled pilot trial to examine the impact of inhaled budesonide on non-ventilated infants.

The study objectives, in a cohort of very preterm infants with signs of early BPD are: 1) to evaluate the effect of aerosolized budesonide on 'days on supplemental oxygen', and 2) to gain an estimate of the impact on BPD and 3) to assess the safety of the intervention in a small cohort of preterm infants.

This will be a single-center randomized double-blind controlled pilot trial. We will recruit a total of 50 infants born at less than 30 weeks gestation who are on continuous positive airway pressure (CPAP) with fraction of inspired oxygen ≥25% on day 14 of life or later. Inhaled budesonide 1mg (intervention group) or normal saline (placebo) will be administered three times a day until the infants do not need CPAP or supplemental oxygen or reach 36+0/7 weeks corrected gestational age. We will evaluate 'days on supplemental oxygen', BPD, re-intubation rates, days on mechanical ventilation and days on CPAP as well as adverse outcomes.

The prevention of BPD would have a significant positive impact on patient quality of life and medical resource utilization and costs. The study hypothesis is that inhaled budesonide on non-ventilated infants with early signs of BPD will reduce the 'days on supplemental oxygen' indicating a positive effect for the prevention of BPD. The result of this pilot study might also justify and support to proceed to a large confirmatory study to evaluate an effect of the intervention on BPD, in which the estimate of the impact on BPD gained in this pilot trial may be used to calculate a sample size.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous breathing preterm Infants on day 14 to day 42 of age
* Born at < 30 0/7 weeks gestational age
* Requiring FiO2 ≥ 25% on CPAP including biphasic CPAP or high flow nasal canula

Exclusion Criteria:

* Presence of chromosomal defects or major congenital anomalies
* Presence of severe infections including sepsis, meningitis, pneumonia, systemic fungal infections
* History of administration of systemic corticosteroids for pulmonary problems, not including that for hypotension

Ages: 14 Days to 42 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Total days on supplemental oxygen from birth to discharge | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks

SECONDARY OUTCOMES:
Bronchopulmonary dysplasia | At 36+0/7 weeks corrected gestational age
  Bronchopulmonary dysplasia is defined as supplemental oxygen use at 36+0/7 weeks corrected gestational age
Mortality (all causes) | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
Death or bronchopulmonary dysplasia | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
Days on supplement oxygen after the study enrollment | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
Days on continuous positive airway pressure (CPAP) | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  Support with continuous positive airway pressure, including use of biphasic CPAP and high flow nasal canula (>= 1L/minutes).
Days with significant apneas | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  Significant apneas with more than 12 episodes requiring stimulation or more than one episode requiring mask-bagging in a six hour period
Culture proven sepsis | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
Gastrointestinal bleeding | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
Persistent hyperglycemia | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  blood glucose > 10mmol/L more than twice in one day
Hypertension | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  blood pressure ≥ 95th percentile for infant's gestational and postnatal ages
Salivary cortisol level | 2 weeks after the study entry and at the first follow up visit at 6 week's corrected age
Postnatal growth | at 36 weeks corrected gestational age and at first follow-up visit at 6 weeks' corrected age
  Weight, Head Circumference and Length
Patent ductus arteriosus | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  PDA diagnosed clinically or by echocardiography

OTHER OUTCOMES:
Intraventricular hemorrhage | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  Any grade of intraventricular hemorrhage as assessed on cranial ultrasound
Periventricular leukomalacia | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  Cystic periventricular leukomalacia as assessed by cranial ultrasound
Retinopathy of prematurity | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  Stage 3 or 4 or surgery as determined from ophthalmological examination
Necrotizing enterocolitis | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  Bell's stage 2 or higher

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dunn, M.D., Principal Investigator — Staff Neonatologist; Tetsuya Isayama, M.D., Principal Investigator — Clinical Fellow
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No